CLINICAL TRIAL: NCT07185828
Title: Informing Low-acuity Emergency Department Patients of Non-emergent Healthcare Resources Following Discharge to Decrease Emergency Department Utilization (2)
Brief Title: Informing Low-acuity Emergency Department Patients of Non-emergent Resources (2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0183-2
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Emergency Service, Hospital; Behavior Change Interventions
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Masking Description: Patients will be aware of their own messages but not of messages sent to other patients or in other arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This arm will receive no intervention outside of usual care.
- Contact your PCP (Experimental): Intervention content emphasizes contacting a primary care provider (content will vary slightly based on whether the patient has a Geisinger PCP)
  Interventions: Behavioral: Contact your PCP
- Use Intelligent Triage (Experimental): Intervention content emphasizes using Intelligent Triage to assess symptoms.
  Interventions: Behavioral: Use Intelligent Triage

INTERVENTIONS:
Behavioral: Contact your PCP — Text messages will be sent and discharge paperwork will be modified to encourage contacting a primary care provider.
  Arms: Contact your PCP
Behavioral: Use Intelligent Triage — Text messages will be sent and discharge paperwork will be modified to encourage using Intelligent Triage.
  Arms: Use Intelligent Triage

SUMMARY:
The goal of this campaign is to reduce unnecessary visits to a Geisinger emergency department (ED). In this campaign, patients will be assigned to receive or not receive outreach following ED discharge with a low-acuity visit designation. Outreach will occur via a text message the day after discharge from the ED as well as information added to the patient's after visit summary (AVS). Depending on the assigned condition, it will include calls to see their primary care provider (PCP) or use an Intelligent Triage tool. The study will assess whether ED use within the following 120 days differs across patients in different outreach conditions (current standard practice vs contact your PCP vs use Intelligent Triage). It will also examine whether patients follow through on the message-specific calls to action differently across conditions.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Geisinger ED visit rated as low acuity (L4 or L5)
* Discharged from Geisinger ED in past 24 hours

Exclusion Criteria:

* Cannot be contacted via the communication modality being used in the study (i.e., SMS), due to insufficient/missing contact information in the EHR or because the patient opted out
* Admitted to hospital
* Already included in intervention in past 365 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8286 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Return to Geisinger ED | within 120 days following day of discharge
  ED visit (yes/no)

OTHER OUTCOMES:
PCP appointment made | within 60 days following day of discharge
  PCP appointment made (yes/no)
PCP visit | within 60 days following day of discharge
  PCP appointment attended (yes/no)
Telehealth appointment made | within 60 days following day of discharge
  Telehealth appointment made (yes/no)
Telehealth appointment attended | within 60 days following day of discharge
  Telehealth appointment attended (yes/no)
Call made to PCP | within 60 days following day of discharge
  Record of patient call to PCP (yes/no)
Urgent care visit | within 60 days following day of discharge
  Urgent care appointment attended (yes/no)
Used Intelligent Triage | within 60 days following day of discharge
  Used the Intelligent Triage tool (yes/no)
Any of the suggested actions taken | within 60 days following day of discharge
  PCP called or visited, telehealth appointment attended, or PCP or telehealth appointment made, or Intelligent Triage tool used (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT07185828/Prot_SAP_000.pdf